CLINICAL TRIAL: NCT07078994
Title: A Randomized Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of BCD-261 in Subjects With Moderate to Severe Active Crohn's Disease
Brief Title: Clinical Study of the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of BCD-261 in Subjects With Moderate to Severe Active Crohn's Disease
Acronym: COMANDOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-261-2
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease (CD)
Keywords: biologics; Crohn's disease; monoclonal antibodies; TL1A
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BCD-261, medium dose induction/ low dose maintenance regimens (Experimental): Subjects in this arm will receive a medium dose of the BCD-261 during the induction regimen (Weeks 0-12), followed by a transition to a maintenance regimen with a low dose of the BCD-261
  Interventions: Biological: anti-TL1A monoclonal antibody, low dose; Biological: anti-TL1A monoclonal antibody, medium dose
- BCD-261, medium dose induction/ medium dose maintenance regimens (Experimental): Subjects in this arm will receive a medium dose of the BCD261 during both the induction phase (Weeks 0-12) and the maintenance regimen
  Interventions: Biological: anti-TL1A monoclonal antibody, medium dose
- BCD-261, high dose induction/ medium dose maintenance regimens (Experimental): Subjects in this arm will receive a high dose of the BCD-261 during the induction regimen (Weeks 0-12), followed by a transition to a maintenance regimen with a medium dose of the BCD-261
  Interventions: Biological: anti-TL1A monoclonal antibody, medium dose; Biological: anti-TL1A monoclonal antibody, high dose
- BCD-261, high dose induction/ high dose maintenance regimens (Experimental): Subjects in this arm will receive a high dose of the BCD261 during both the induction phase (Weeks 0-12) and the maintenance regimen
  Interventions: Biological: anti-TL1A monoclonal antibody, high dose
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo till the assessment of the primary endpoint and then will be switched to BCD-261medium studied dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: anti-TL1A monoclonal antibody, low dose — injection
  Arms: BCD-261, medium dose induction/ low dose maintenance regimens
Biological: anti-TL1A monoclonal antibody, medium dose — injection
  Arms: BCD-261, high dose induction/ medium dose maintenance regimens; BCD-261, medium dose induction/ low dose maintenance regimens; BCD-261, medium dose induction/ medium dose maintenance regimens
Biological: anti-TL1A monoclonal antibody, high dose — injection
  Arms: BCD-261, high dose induction/ high dose maintenance regimens; BCD-261, high dose induction/ medium dose maintenance regimens
Other: Placebo — injection
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics and immunogenicity of study drug (BCD-261) in comparison with placebo and to characterize the dose-response relationship in patients with moderate to severe active Crohn's Disease. The study will be conducted in a population of male and female subjects ≥18 years and ≤75 years with moderate to severe active Crohn's Disease and an inadequate response to prior treatment with glucocorticoids, immunosuppressants, or biologics/targeted immunosuppressants.

DETAILED DESCRIPTION:
Subjects meeting the eligibility criteria will be randomized in 5 groups to receive one of four studied dosage regimens of BCD-261 or placebo. The study groups will differ in drug dosages of BCD-261 (low, medium, high) during the induction and maintenance periods of therapy. After the primary endpoint assessment subjects in placebo group will be switched to BCD-261 medium studied dose.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of Crohn's disease involving the terminal ileum or colon (types L1-L3 according to the Montreal classification), established ≥3 months prior to signing the informed consent form and confirmed by endoscopic findings.
2. Moderate to severe active Crohn's disease, manifested by the following signs:

(1) Crohn's Disease Activity Index (CDAI) ≥220 and ≤450 points.

(2) Simple Endoscopic Score for Crohn's Disease (SES-CD) ≥6 points or ≥4 points for the disease form with isolated involvement of the ileum (according to central independent review).

3. Inadequate response to therapy according to the investigator's assessment, manifested by at least one of the following signs:

1. Persistent symptoms of disease activity despite treatment with at least one course of glucocorticoids including prednisolone at a dose of ≥40 mg/day or equivalent or budesonide ≥9 mg/day or equivalent for at least 2 weeks with oral administration (at least 1 week with intravenous administration at a dose equivalent to oral prednisolone ≥40 mg/day).
2. Steroid dependence manifested by an increase in disease activity after initial improvement, with a decrease in the dose of glucocorticoids below the dose equivalent to 10 mg of oral prednisolone per day, within 3 months from the beginning of treatment, or a relapse of the disease within 3 months after the end of glucocorticoid use.
3. Persistent symptoms of disease activity despite treatment with at least one course of immunosuppressants (azathioprine at a dose of ≥2.0 mg/kg and/or 6-mercaptopurine at a dose of ≥1.0 mg/kg and/or methotrexate at a dose of ≥15.0 mg/week) for ≥12 weeks, or in response to another treatment regimen with these drugs according to a regional standard of care.
4. Primary lack of response to therapy with TNFa inhibitors and/or anti-integrins, and/or IL-12/23 inhibitors, and/or targeted immunosuppressors (upadacitinib), defined as the persistence of symptoms of disease activity despite at least one course of induction of remission according to a treatment scheme approved by the regional standard.
5. Loss of response to therapy with TNFa inhibitors and/or anti-integrins, and/or IL-12/23 inhibitors, and/or targeted immunosuppressors (upadacitinib), defined as the appearance of symptoms of disease activity after initial improvement as a result of treatment with at least one course of induction of remission and at least one course of maintenance of remission according to a treatment scheme approved by the regional standard.
6. A history of intolerance to glucocorticoid therapy and/or immunosuppressors (azathioprine, 6-mercaptopurine, methotrexate) and/or biologic therapies (TNFα inhibitors, anti-integrins, IL-12/23 inhibitors) and/or targeted immunosuppressors (upadacitinib), as determined by the treating physician.

4. Maintaining a stable dose of concomitant medications for ≥2 weeks prior to signing the ICF and in the screening period for glucocorticoids and for ≥4 weeks prior to signing the

ICF and in the screening period for immunosuppressants (azathioprine, 6-mercaptopurine, methotrexate).

Exclusion Criteria:

1. A history of or current at the time of signing the ICF ulcerative colitis, unspecified colitis, ischemic colitis, radiation colitis, microscopic colitis, complicated form of diverticular disease.
2. A history of primary sclerosing cholangitis.
3. Presence of active intra-abdominal or perianal abscess at the time of signing the ICF.
4. Presence of an endoscopically obstructed stricture/stenosis of the intestine at the time of signing the ICF.
5. A history of toxic megacolon, intestinal obstruction, intestinal perforation (except for those caused by injury or appendicitis).
6. A history of dysplasia in any part of the gastrointestinal tract at the time of signing the ICF.
7. Previous resections of the small intestine with a total length of resected segments >100 cm and/or resection of >2 segments of the large intestine (ascending colon (including the cecum), transverse colon, descending colon (including the sigmoid colon), rectum)3.
8. Presence of intestinal stoma or artificial rectum or the need for them.
9. Failure of ≥3 classes of biologics/targeted immunosuppressors (according to INN) with different mechanisms of action (TNFa inhibitors, anti-integrins, IL-12/23 inhibitors, upadacitinib) or ≥4 biologics/targeted immunosuppressants (according to INN), regardless of the mechanism of actio

   * Use of any of the indicated therapies within the specified time frame or need for therapy with these drugs during the study period:

     1. Use of TNFa inhibitors within 8 weeks prior to signing the ICF or during the screening period.
     2. Use of anti-integrins or IL-12/23 inhibitors within 12 weeks before signing the ICF or during the screening period.
     3. Use of Janus kinase inhibitors (upadacitinib) within 2 weeks prior to signing the ICF or during the screening period.
     4. Use of oral glucocorticoids at a dose equivalent to prednisone >20 mg/day or budesonide >9 mg/day or rectal administration of glucocorticoids at any dose within 2 weeks prior to signing the ICF or during the screening period or parenteral administration of glucocorticoids at any dose within 4 weeks prior to signing the ICF or during the screening period.
     5. Use of immunosuppressants not included in the approved therapy (tacrolimus, cyclosporine, mycophenolate mofetil, rapamycin, leflunomide, penicillamine, etc.) within 4 weeks before signing the ICF or during the screening period.
     6. Long-term regular use of non-steroidal anti-inflammatory drugs (≥3 times a week for ≥6 weeks) for 2 weeks prior to signing the ICF.
     7. Use of any other investigational drugs in other clinical trials at the time of signing the ICF or less than 8 weeks or 5 half-lives (whichever is longer) before the date of signing the ICF or during screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved clinical remission | week 14
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) score of <150
Proportion of subjects who achieved an endoscopic response | week 14
  Proportion of subjects with ≥50% reduction Simple Endoscopic Score for Crohn's Disease (SES-CD) from the baseline

SECONDARY OUTCOMES:
Proportion of subjects who achieved clinical remission | week 24
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) score of <150

OTHER OUTCOMES:
Proportion of subjects who achieved a clinical response | weeks 14, 24, 52, and 100
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) score reduction ≥100-point from baseline
Proportion of subjects who achieved clinical remission | weeks 52, 100
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) of <150
Proportion of subjects who achieved clinical remission | weeks 24, 52, and 100
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) score of <150 points among subjects who had achieved a clinical response, defined as a ≥100-point reduction from baseline in the CDAI score at Week 14
Proportion of subjects who achieved clinical remission | weeks 52 and 100
  Proportion of subjects with Crohn's Disease Activity Index (CDAI) score of <150 points without the use of glucocorticoids (for at least 12 weeks) among subjects who were initially receiving glucocorticoid therapy
Proportion of subjects who achieved a clinical response | weeks 14, 24, 52, and 100
  Proportion of subjects with ≥50% reduction from baseline on the PRO2 scale (abdominal pain, frequency of loose/very soft stools)
Proportion of subjects who achieved clinical remission | weeks 14, 24, 52, and 100
  Proportion of subjects with abdominal pain intensity score of ≤1 and a frequency of loose/very soft stools score of ≤3 on the PRO2 scale, but not higher than baseline for each parameter
Proportion of subjects who achieved an endoscopic response | weeks 24, 52, 100
  Proportion of subjects with the Simple Endoscopic Score for Crohn's Disease (SES-CD) reduction ≥50% from baseline
Proportion of subjects who achieved endoscopic remission | weeks 14, 24, 52, and 100
  Proportion of subjects with SES-CD ≤4 points, with no more than 1 point for each category
Proportion of subjects who achieved an endoscopic response | Weeks 24, 52, and 100,
  Proportion of subjects with the Simple Endoscopic Score for Crohn's Disease (SES-CD) reduction ≥50% from baseline among subjects who had achieved a clinical response, defined as a ≥100-point reduction from baseline in the CDAI score at Week 14
Change in the fecal calprotectin level from the baseline | Weeks 14, 24, 52, 100
Change in the highly sensitive C-reactive protein level from the baseline | weeks 14, 24, 52, 100
Changes in the proportion of subjects with extra-intestinal manifestations from the baseline | weeks 14, 24, 52, 100

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, Study Director — Director of Clinical Development Department, BIOCAD
Locations (19):
- Russia (19):
  - LLC Medical Center "ASTRA", Barnaul, Altayskiy Kray
  - Republican Clinical Hospital named after G.G. Kuvatov, Ufa, Bashkortostan Republic
  - State Institution of Healthcare of the Moscow Region "Moscow Regional Research Clinical Institute named after M.F. Vladimirsky", Moscow, Moscow
  - Llc "Novosibirsk Gastrocenter", Novosibirsk, Novosibirsk Oblast
  - Federal State Educational Institution of Higher Education "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don, Rostov Oblast
  - LLC "Research Center Eco-Safety", Saint Petersburg, Sankt-Peterburg
  - State Autonomous Institution of Healthcare "Republican Clinical Hospital of the Ministry of Healthcare of the Republic of Tatarstan", Kazan', Tatarstan Republic
  - "South Ural State Medical University" of the Ministry of Health of the Russian Federation, Chelyabinsk
  - Federal Siberian Scientific and Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk
  - Regional State Healthcare Institution "Regional Clinical Hospital, Krasnoyarsk
  - Llc "Olla-Med", Moscow
  - Moscow Clinical Scientific and Practical Center named after A.S. Loginov of the Moscow City Health Department, Moscow
  - State Healthcare Institution of the City of Moscow "V.M. Buyanov City Clinical Hospital of the Moscow City Healthcare Department", Moscow
  - Branch of the LLC "Hadassah Medical LTD", Moscow
  - Federal State Educational Institution of Higher Education "North-West State Medical University named after I.I. Mechnikov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Saint Petersburg State Healthcare Institution "City Hospital of the Holy Martyr Elizabeth", Saint Petersburg
  - Federal State Educational Institution of Higher Education "First Saint Petersburg State Medical University named after Academician I.P. Pavlov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - State Healthcare Institution Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - State Healthcare Institution "Primorsky Regional Clinical Hospital No. 1", Vladivostok

IPD SHARING:
Plan to Share IPD: No